CLINICAL TRIAL: NCT00812942
Title: Participation to Colorectal Cancer Screening With Faecal Occult Blood Test and Colonoscopy: an Italian, Multicenter, Randomized Population Study
Brief Title: Participation to Colorectal Cancer Screening With Fecal Occult Blood Test and Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Superiore di Sanità (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1
Record Dates: First submitted 2008-12-18; First posted 2008-12-22 (Estimated); Last update posted 2008-12-22 (Estimated); Status verified 2008-12

CONDITIONS: Colorectal Cancer
Keywords: average-risk subjects for
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- fobt (Active Comparator): faecal occult blood test
  Interventions: Procedure: faecal test
- colonoscopy (Active Comparator): colonoscopy screening
  Interventions: Procedure: colonoscopy

INTERVENTIONS:
Procedure: colonoscopy — colonoscopy screening
  Arms: colonoscopy
Procedure: faecal test — faecal occult blood test for screening
  Arms: fobt

SUMMARY:
Adherence rate to screening colonoscopy (TC) in the average-risk general population is still unclear. Aim of this study was to compare the uptake of TC screening with that of fecal occult blood (FOBT) in the general population of different Italian areas.

DETAILED DESCRIPTION:
A nationwide, population-based, multicenter, randomized trial comparing attendance to TC with that to FOBT was performed. Sixty-four general practitioners (GPs), overall including in their lists 9,889 average-risk subjects aged 55-64 years, were randomized between TC and FOBT screening programs. Eligible subjects were mailed a personal invitation letter co-signed by their GP and the coordinator of the area-reference GI centre. Attendance rate and detection rate for advanced neoplasia (colorectal cancer, adenoma >10 mm or with villous histology or high-grade dysplasia) for each arm of the study were assessed.

ELIGIBILITY:
Inclusion Criteria:

* asymptomatic 55-64 years subjects

Exclusion Criteria:

* already studied for colorectal cancer, severe comorbidities

Ages: 55 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9889 (Actual)
Dates: Start 2003-11; Primary Completion 2005-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Participation to colorectal cancer screening

CONTACTS AND LOCATIONS:
Locations (1):
- IIstituto Nazionale Tumori Regina Elena, Rome, Italy